CLINICAL TRIAL: NCT07031713
Title: A Clinical Study Exploring the Safety, Efficacy and Cell Metabolic Dynamics of Universal CD19 / 20 Car-t Cell Injection in Moderate to Severe Refractory Systemic Lupus Erythematosus
Brief Title: Safety, Efficacy and Cellular Metabolic Dynamics of ct1192 in Patients With Moderate to Severe Refractory SLE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Qiubai Li, Director, Head of Department of Rheumatology and Immunology, Principal Investigator, Professor, Wuhan Union Hospital, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT1192-CG11003_01
Record Dates: First submitted 2025-06-04; First posted 2025-06-22 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-06

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT1192 CAR-T cells Injection (Experimental): CT1192 cells infusion
  Interventions: Biological: CAR-T Therapy

INTERVENTIONS:
Biological: CAR-T Therapy — CT1192 cells infusion

SUMMARY:
A clinical study to explore the safety, efficacy and cell metabolic kinetics of universal CD19/20 car-t cell injection in moderate to severe refractory systemic lupus erythematosus.

This study is a single arm, open, exploratory dose increasing clinical study, which aims to evaluate the safety, efficacy and cell metabolic dynamics of ct1192 cells in patients with SLE.

DETAILED DESCRIPTION:
The study was divided into dose increasing stage and dose expanding stage. dose escalation phase Three dose levels are tentatively determined for dose escalation: 3.0 × 108, 4.5 × 108 and 6.0 × 108 car-cd19/CD20+T cells. It is estimated that the target toxicity probability of the maximum tolerated dose is 30%, and about 12 participants are planned to be enrolled, and the number of enrolled patients in each dose group is subject to the actual situation. During the test, the researchers and partners will jointly negotiate whether to increase or decrease the dose, whether to increase to the set maximum dose group or produce the maximum available cell volume, and whether to increase the exploration of new dose level within the explored dose range (allowed to be conducted when the dose is increased or decreased) according to the participants' cell metabolism characteristics, safety, tolerance and preliminary effectiveness data, so as to determine the possible recommended therapeutic dose (RD).

The DLT observation period is 28 days after the first infusion. If the treatment needs to be withdrawn before 28 days after the infusion due to disease progression or other reasons, no obvious car-t cell expansion is detected or car-t treatment is invalid, and the DLT related AE events determined by the researcher may not be related to the product, the DLT observation period can be completed before. During each dose increase, if there is a safety risk that needs to be discussed, the researchers and partners can make a dose increase/stability/decrease decision according to the safety and tolerance of participants and the metabolic kinetics of ct1192 cells. In the same dose group, the first participant had no significant safety risk 14 days after the completion of cell infusion, and subsequent participants could only carry out cell infusion.

dose expansion phase One or more dose groups may be selected for dose expansion according to the results of the dose increasing stage to further explore the efficacy and safety in SLE patients. Each dose group and each queue plan to include up to 9 cases, and the specific number of patients in the group is subject to the actual number. DLT will not be observed in the dose expansion phase, and other research processes are the same as the dose increment phase. Researchers and collaborators will continue to monitor the safety data of the whole dose expansion phase and make decisions on admission and exit when necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the EULAR/ACR 2019 SLE classification criteria, with a medical history of ≥ 6 months;
2. Voluntarily sign the Informed Consent Form (ICF); When signing the ICF, the age range is between 18 and 60 years old (including 18 and 60 years old), with no gender restrictions;
3. No systemic active infections (such as infectious pneumonia or tuberculosis) within the first 2 weeks of screening;
4. Women with fertility (defined as all physiologically capable women) must agree to use effective contraceptive methods from at least 28 days prior to the start of vaginal discharge until 1 year after CT1192 infusion. Egg donation is strictly prohibited within 1 year after receiving the study treatment infusion during the study period. Male partners with fertility must agree to use effective barrier contraception methods from the start of vaginal discharge until 1 year after CT1192 infusion, and should not donate semen or sperm throughout the entire study period;
5. Women with fertility must have a negative serum β - human chorionic gonadotropin (β - hCG) test result within 48 hours prior to screening and gonorrhea treatment.
6. Prior to screening, patients must have received a combination of glucocorticoids and immunosuppressants (including cyclophosphamide, mycophenolate mofetil, tacrolimus, methotrexate, cyclosporine, leflunomide) and/or biologics for at least 3 months, with a stable dose for at least 2 weeks and the disease still active. During screening, oral steroids must meet the following requirements:

If hormone therapy is used alone, prednisone (or equivalent medication) should be ≥ 7.5 mg/day; When used in combination with immunosuppressants and/or biologics, there is no minimum daily dose requirement for hormones; 7. Positive for anti nuclear antibodies, anti ds DNA antibodies, and/or anti Smith antibodies during screening; 8. During the screening period, if the SLEDAI-2K score is ≥ 7 points, or if there is significant organ dysfunction, such as severe immune thrombocytopenia or lupus nephritis (histologically diagnosed as active nephritis type III or IV with or without type V); 9. Active organ involvement during screening (including kidneys, heart and lungs, musculoskeletal system, blood system, blood vessels, etc.; skin and mucosal involvement alone cannot be included); 10. Adequate organ function:

1. Renal function: defined as a creatinine clearance rate (Cockcroft Gault) calculated without hydration assistance of ≥ 50 mL/min;
2. Bone marrow function: defined as neutrophil count (ANC) ≥ 1.0 × 109/L and hemoglobin (Hb) ≥ 60 g/L. Blood transfusions and growth factors must not be used to meet these requirements within 7 days prior to eligibility screening;
3. Liver function: defined as alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2 x upper limit of normal (ULN), total bilirubin ≤ 2 x upper limit of normal (ULN)
4. Coagulation function: defined as International Normalized Ratio (INR) or Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN;
5. Pulmonary function: Blood oxygen saturation (SpO2) ≥ 92% in indoor air (measured by pulse oximeter);
6. Cardiac function: defined as a left ventricular ejection fraction (LVEF) of ≥ 50% evaluated by echocardiography (ECHO) within the first 8 weeks of screening.

Exclusion Criteria:

1. Patients with severe lupus nephritis within the first 2 months of screening need to undergo hemodialysis or receive prednisone ≥ 100 mg/d or equivalent hormone therapy for ≥ 14 days;
2. Have undergone plasma exchange, plasma separation, hemodialysis within 30 days prior to screening, or have had lupus crisis within 30 days prior to screening;
3. Individuals with a history of ≥ grade 2 bleeding or requiring long-term anticoagulant therapy within the 30 days prior to screening;
4. Screening for a history of any of the following cardiovascular diseases within the previous 30 days: Grade III or IV heart failure defined by the New York Heart Association (NYHA), myocardial infarction, unstable angina, uncontrolled or symptomatic atrial arrhythmias, any ventricular arrhythmias, or other clinically significant heart diseases;
5. Prior to screening, central nervous system manifestations caused by lupus, including but not limited to lupus headache, epileptic seizures, cognitive impairment, impaired intellectual function, visual impairment, etc;
6. Individuals with central nervous system diseases prior to screening include but are not limited to: cerebrovascular accidents, encephalitis, epilepsy, seizures/convulsions, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar diseases, central nervous system vasculitis, cognitive dysfunction, organic brain syndrome, or psychiatric disorders;
7. No systemic active infections, including but not limited to active tuberculosis, within 2 weeks prior to screening;
8. Previously received CAR-T cell or other genetically modified T cell therapy, or have a history of major organ transplantation (such as heart, lung, kidney, liver) or hematopoietic stem cell/bone marrow transplantation;
9. Allergic or intolerant reactions to Qinglin drugs, tocilizumab, or life-threatening allergic reactions, hypersensitivity reactions, or intolerance to CT1192 preparations or their excipients (including dimethyl sulfoxide (DMSO)), or previous history of other severe allergies such as anaphylactic shock;
10. Screening for drugs targeting B cells, such as rituximab, that have been used within the previous 6 months;
11. Within the 12 weeks prior to screening, other biologics such as taceptil and belimumab have been used for treatment;
12. Hormone use ≥ 10 mg/day of prednisone (or equivalent) within 2 weeks prior to CT1192 infusion, with the use of physiological substitutes, topical and inhaled steroids allowed;
13. Received immunosuppressive agents that affect T cells (mycophenolate mofetil, methotrexate, cyclosporine, azathioprine, leflunomide, tacrolimus) within 2 weeks prior to CT1192 infusion;
14. Have received JAK inhibitors (tofacitinib, baritinib tablets, lukatinib, etc.) within 2 weeks prior to CT1192 infusion;
15. Have received attenuated live vaccine, inactivated vaccine or RNA vaccine within one month before screening;
16. Suffering from malignant tumors within 2 years prior to signing the ICF. Except for the following situations: non melanoma skin cancer that has undergone radical treatment, local prostate cancer, cervical carcinoma in situ confirmed by biopsy or squamous intraepithelial lesions detected by cervical smear, and breast carcinoma in situ that has been completely removed;
17. If a major surgery has been performed within 4 weeks prior to signing the informed consent form, or if a major surgery is planned during the study period, the researcher believes that it would pose unacceptable risks to the participants; During screening, there may be HIV, syphilis infection, active hepatitis B virus infection (HBsAg positive and HBV-DNA above the detection limit), or active hepatitis C virus infection (HCV antibody and HCV-RNA positive);

19. Participate in other clinical studies within the first 3 months of screening or still within the five half lives after the last medication; 20. Merge major chronic diseases that have not been controlled and researchers believe may increase the risk for participants; 21. If there is a history or evidence of suicidal thoughts within the previous 6 months, or any suicidal behavior within the previous 12 months, the researcher believes that there is a significant risk of suicide; 22. Pregnant or lactating women; According to the researcher's assessment, participants have poor compliance, are unable or unwilling to comply with the requirements of the research protocol, or are not suitable to participate in this clinical study for other reasons.

5.5 Pre cleaning standard Before clearing, the following assessment needs to be completed. If the participant meets the following criteria, clearing can be performed. Otherwise, clearing cannot be performed or may need to be delayed.

1. Not using immunosuppressants in the week before Qinglin treatment;
2. Female participants with fertility potential who undergo pregnancy studies within 24 hours prior to the clearance of gonorrhea and have negative results;
3. Blood oxygen saturation ≥ 92% (under non auxiliary oxygen supply conditions);
4. Inactive or uncontrollable systemic infection; The use of anti infective drugs within 7 days before clearing gonorrhea must be reviewed by a medical inspector;
5. No signs of CNS disease or abnormal neurological examination results with clinical significance;
6. Serious abnormalities in heart, lung, liver, kidney function, and endocrine disorders, including but not limited to: newly developed arrhythmias or heart failure that cannot be controlled by medication; Hypotension requiring the use of vasopressors; Bacterial, fungal, or viral infections with increased activity/progression determined by researchers;
7. Researchers assess that participants are unable to comply with the requirements of the study protocol or are not suitable to continue the study in other situations.

If a participant shows obvious abnormalities such as symptoms, signs, or test results during or after clearing the lymphatic system, the researcher must communicate with the cooperating medical monitor to discuss whether the participant is suitable to continue receiving CT1192 cell infusion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ct1192 in participants with moderate to severe refractory SLE | Within 28 days after infusion for DLT, within 180 days after infusion fOr AE/SAEwithin 12 months after infusion for AESl
  The incidence and severity of dose limiting toxicity (DLT), adverse events (AE), serious adverse events (SAE), and AESI (adverse events of particular concern)
Evaluate the maximum tolerable dose (MTD) and/or dose range of ct1192 | After medication to day 28
  Ct1192 MTD and/or dose range

SECONDARY OUTCOMES:
Proportion of participants with SLE responder index (sri-4) | 1, 3, 6, 9 and 12 months after drug use
  Preliminary evaluation of the efficacy of ct1192 in the treatment of moderate to severe refractory SLE.Proportion of participants who reached SLE responder index (sri-4) at 6 months and other time points (1, 3, 9 and 12 months after medication)
Proportion of participants with low lupus disease activity status (lldas) | 1, 3, 6, 9 and 12 months after drug use
  To evaluate the efficacy of ct1192 in the treatment of moderate to severe refractory SLE. The proportion of participants who reached lupus low disease activity status (lldas) at 6 months and other time points (1, 3, 9 and 12 months after medication).
Proportion of participants achieving disease remission (doris) | 1, 3, 6, 9 and 12 months after drug use
  To evaluate the efficacy of ct1192 in the treatment of moderate to severe refractory SLE. The proportion of participants who achieved disease remission (doris) at 6 months and other time points (1, 3, 9 and 12 months after medication).
Changes of SLE disease activity index (sledai-2k) score from baseline after medication | 1, 3, 6, 9 and 12 months after drug use
  To evaluate the efficacy of ct1192 in the treatment of moderate to severe refractory SLE. The SLE disease activity index (sledai-2k) scores at 6 months and other time points (1, 3, 9 and 12 months) after treatment were changed from baseline.
After treatment, the SLE disease activity index (Selena - SLEDAI) score changed from baseline | 1, 3, 6, 9 and 12 months after drug use
  To evaluate the efficacy of ct1192 in the treatment of moderate to severe refractory SLE. The SLE disease activity index (Selena - SLEDAI) scores at 6 months and other time points (1, 3, 9 and 12 months) after treatment were changed from baseline.
After treatment, the index of lupus erythematosus assessment group (bilag-2004) changed from baseline | 1, 3, 6, 9 and 12 months after drug use
  Preliminary evaluation of the effectiveness of CT1192 for moderate to severe refractory SLE. Changes in the British Islet Lupus Assessment Group Index (BILAG-2004) compared to baseline at 6 months and other time points (1, 3, 9, and 12 months) after medication.
The SLE activity score (sle-das) changed from baseline after treatment | 1, 3, 6, 9 and 12 months after drug use
  Preliminary evaluation of the effectiveness of CT1192 for moderate to severe refractory SLE. Changes in SLE Disease Activity Score (SLE-DAS) compared to baseline at 6 months and other time points (1, 3, 9, and 12 months) after medication.
Changes in clinicians' overall judgment (PGA) score from baseline after medication | 1, 3, 6, 9 and 12 months after drug use
  Preliminary evaluation of the effectiveness of CT1192 for moderate to severe refractory SLE. The overall assessment (PGA) score of clinical physicians changed from baseline at 6 months and other time points (1, 3, 9, and 12 months) after medication.
Proportion of patients without other SLE therapy after medication | 1, 3, 6, 9 and 12 months after drug use
  Preliminary evaluation of the effectiveness of CT1192 for moderate to severe refractory SLE. The proportion of patients without other SLE therapies at 1, 3, 6, 9, and 12 months after medication.
Changes in immunoglobulin (IgG, IgM, IgA) levels during medication | 1, 3, 6, 9 and 12 months after drug use
  Preliminary evaluation of the effectiveness of CT1192 for moderate to severe refractory SLE. Changes in immunoglobulin (IgG, IgM, IgA) levels at 1, 3, 6, 9, and 12 months after medication.
The changes of serum markers (anti DS DNA antibody, anti Smith antibody, antinuclear antibody Ana, complement C3) of SLE after treatment | 1, 3, 6, 9 and 12 months after drug use
  Preliminary evaluation of the effectiveness of CT1192 for moderate to severe refractory SLE. Changes in serum markers of SLE disease (anti ds DNA antibody, anti Smith antibody, anti nuclear antibody ANA, complement C3) levels at 1, 3, 6, 9, and 12 months after medication.
The change value of post medication Health Assessment Questionnaire Disability Index (HAQ-DI) from baseline | 1, 3, 6, 9 and 12 months after drug use
  Preliminary evaluation of the effectiveness of CT1192 for moderate to severe refractory SLE. Changes in Health Assessment Questionnaire Disability Index (HAQ-DI) from baseline at 1, 3, 6, 9, and 12 months after medication.
Copy number and duration of ct1192 gene in blood | Within 1 year after CAR-T cell infusion
  Objective to evaluate the cell kinetics of ct1192 in SLE participants, and to observe the level and duration of ct1192 gene copy number in blood.
Changes of B cell functional subsets (initial B cells, memory B cells, plasma cells) after ct1192 infusion | Within 1 year after CAR-T cell infusion
  Evaluate the efficacy (PD) characteristics of CT1192 in SLE participants. Changes in the levels of B cell functional subgroups (initial B cells, memory B cells, plasma cells) after CT1192 infusion.
Changes in cytokine levels after CT1192 infusion | Within 1 year after CAR-T cell infusion
  Evaluate the efficacy (PD) characteristics of CT1192 in SLE participants. Changes in cytokine levels after CT1192 infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospita, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No